CLINICAL TRIAL: NCT03341871
Title: Glecaprevir/Pibrentasvir Drug Use Results Survey in Patients Infected With Hepatitis C Virus Genotype 1-6
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-570
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: chronic hepatitis C virus (HCV); Genotype; glecaprevir; pibrentasvir; sustained virologic response; chronic hepatitis C virus genotype 1; chronic hepatitis C virus genotype 2; chronic hepatitis C virus genotype 3; chronic hepatitis C virus genotype 4; chronic hepatitis C virus genotype 5; chronic hepatitis C virus genotype 6
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HCV Genotypes 1, 2, 3, 4, 5, or 6 participants: Participants receiving combination therapy with the glecaprevir plus pibrentasvir (GLE/PIB) regimen according to the current local label.

SUMMARY:
This multi-center, post-marketing, observational study evaluates the real world safety and effectiveness of glecaprevir plus pibrentasvir use in participants infected with the hepatitis C virus genotype 1 - 6.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C virus infection and administering glecaprevir plus pibrentasvir.

Exclusion Criteria:

* Patients previously treated with glecaprevir plus pibrentasvir.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japan patients infected with hepatitis C virus and treating with glecaprevir plus pibrentasvir per approved Japan label.
Sampling Method: Non-Probability Sample
Enrollment: 1095 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Sustained Virological Response 12 Weeks Post-treatment (SVR12) | 12 weeks after last dose of drug
  SVR12 defined as the hepatitis C virus (HCV) ribonucleic acid (RNA) level < the lower limit of quantification (LLOQ) 12 weeks after the last dose of Glecaprevir plus Pibrentasvir.

SECONDARY OUTCOMES:
Percentage of Participants with Post-treatment Relapse | Up to 24 weeks after last dose of drug
  Post-treatment relapse was defined as confirmed HCV RNA >= LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Percentage of Participants with On-treatment Virologic Failure | Up to 12 weeks after first dose
  On-treatment virologic failure was defined as HCV RNA levels reach < LLOQ during treatment then increase to >= LLOQ during treatment, or confirmed increase of > 1 log10 IU/mL above the lowest value post-baseline HCV RNA during treatment.
Percentage of Participants Achieving SVR4 | 4 weeks after last dose
  SVR4 defined as defined as the HCV RNA level < LLOQ 4 weeks after the last dose of Glecaprevir plus Pibrentasvir.
Percentage of Participants Achieving SVR8 | 8 weeks after last dose of drug
  SVR8 defined as defined as the HCV RNA level < LLOQ 8 weeks after the last dose of Glecaprevir plus Pibrentasvir.
Percentage of Participants Achieving SVR24 | 24 weeks after last dose of drug
  SVR24 defined as the HCV RNA level < LLOQ 24 weeks after the last dose of Glecaprevir plus Pibrentasvir.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (1):
- Abbvie Japan /ID# 161985, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/ombitasvir_dasabuvir_P16-570.pdf